CLINICAL TRIAL: NCT00435305
Title: Antibiotic Concentrations in Serum and Epithelial Lining Fluid Under Continous Infusion
Brief Title: Steady State Serum and Epithelial Lining Fluid (ELF) Antibiotics Concentrations Under Continous Infusion
Status: Terminated | Type: Observational
Why Stopped: difficulties by enrolling patients fundings consumed, no staff could be recruited and payed to continue enrolling patients,
Sponsor: University Hospital Tuebingen (Other)
Other Study IDs: 2005-002128-32
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Pneumonia; Bacteremia
Keywords: continuous infusion; epithelial lining fluid; antibiotics; pneumonia; critical illness
MeSH Terms: conditions — Pneumonia; Bacteremia; Critical Illness | interventions — Meropenem; Vancomycin; Linezolid; Piperacillin, Tazobactam Drug Combination; Cefepime; Ceftazidime

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Meropenem
Drug: Vancomycin
Drug: Linezolid
Drug: Piperacillin/Tazobactam
Drug: Cefepim
Drug: Ceftazidim

SUMMARY:
The purpose of our study is to determine the penetration of continuously infused antibiotics at steady state, mainly Meropenem, Vancomycin, Linezolid, Piperacillin/tazobactam and additionally cefepim and ceftazidim, into epithelial lining fluid.

DETAILED DESCRIPTION:
Severe infectious disease may be the cause for admitting a patient to an ICU, but more often they constitute a complication of the intensive care and turn out to be caused by nosocomial pathogens.

Nosocomial infections are associated with a high lethality. The appropriate antibiotic therapy determines in part the outcome of the patients. Especially this antibiotic therapy implicates a number of problems for the physician.

He has to ensure that the chosen antibiotics are effective against the most common and presumed pathogens and that the reached concentrations of antibiotics in plasma and epithelial lining fluid are reliably and permanently above the minimal inhibitory concentration (MIC) for the given pathogens.

All the antibiotics included in our clinical trial are so called "time dependent" antibiotics. They are most effective if there concentrations reach a certain level (MIC) at the infected site (epithelial lining fluid in our study) over the entire period of treatment.

To achieve this aim, many authors already suggested that the continuous infusion might solve the problem of too low antibiotic plasma and ELF levels. Studies about pharmacokinetics of continuous infused antibiotics, which were conducted in healthy volunteers or patients with normal organ function, cannot be assigned to critical ill patients. Rationales for this statement are that data about plasma and tissue levels of antibiotics in critical ill patients are highly influenced by modified volume of distribution, elimination half-life period and impaired tissue perfusion compared to healthy volunteers. These physiological variances implicate that the response to the antibiotic treatment remains doubtful. Under these pathophysiological conditions, data about antibiotics plasma and ELF levels may provide additional information in order to adjust the dosing regime of antibiotics.

Studies conducted in critical ill patients showed that under the circumstances of continuous infused antibiotics, the reached levels in plasma are above the MIC. However there is little data about penetration into ELF of continuous infused antibiotics.

Our study intends to provide data about plasma and ELF levels of continuous infused antibiotics in steady state, determine a penetration coefficient for these antibiotics into ELF and to compare the reached levels in ELF to the MIC.

To demonstrate the efficiency of continuous infused antibiotics, we will conduct quantitative microbiological measurements before and after treatment if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both gender >0 18 years of age
* Patients of an ICU with one or more of the following infections
* Bacteremia. sepsis
* pneumonia
* tracheo-bronchitis
* mechanical ventilation
* stay on the ICU >= 3 days
* indication for bronchoscopy

Exclusion Criteria:

* pregnancy
* allergy against the studied drug
* known resistance of the involved pathogen against the study drug
* simultaneous participation in other studies
* former participation in the present study
* probable stay on the ICU < 3 days
* contra-indication against the study-drug
* contra-indication for bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-11; Study Completion 2007-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Krueger, PHD, Study Chair — Universitätsklinikum Tübingen, Klinik für Anästhesiologie und Intensivmedizin
Locations (1):
- Universitäsklinikum Tübingen, Klinik für Anästhesiologie und Intensivmedizin, Tübingen, Germany